CLINICAL TRIAL: NCT03619031
Title: Effects of Pizza Leavening Process on Postprandial Glucose Response in Patients With Type 1 Diabetes
Brief Title: Pizza Leavening and Postprandial Glycemia in Type 1 Diabetes (LEAVEN)
Acronym: LEAVEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 107/18
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; postprandial glycemia; pizza leavening
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LONG LEAVENING (Experimental): Acute test meal
  Interventions: Other: LONG LEAVENING
- SHORT LEAVENING (Experimental): Acute test meal
  Interventions: Other: SHORT LEAVENING
- TRADITIONAL (Active Comparator): Acute test meal
  Interventions: Other: TRADITIONAL

INTERVENTIONS:
Other: LONG LEAVENING — a long-leavened (60 h) pizza composed of sourdough and a flour mix.
  Arms: LONG LEAVENING
Other: SHORT LEAVENING — a short-leavened (5 h) pizza composed of sourdough and a flour mix.
  Arms: SHORT LEAVENING
Other: TRADITIONAL — a short-leavened (5 h) pizza composed of brewer's yeast and 00 flour.
  Arms: TRADITIONAL

SUMMARY:
The purpose of this study is to compare in patients with type 1 diabetes the postprandial glucose response to the consumption of three types of pizza, obtained with different leavening techniques. The intervention will be preceded by a one-week run-in period during which participants will undergo continuous glucose monitoring (CGM) to optimize basal infusion rate and insulin-to-glycemic load ratio. According to a randomized crossover design, the participants will consume at home at dinner-time in three different days over a 3-week period in random order: 1) a long-leavened pizza, composed of sourdough and a flour mix; 2) a short-leavened pizza, composed of sourdough and a flour mix; 3) a traditional pizza, composed of brewer's yeast and refined wheat flour, used as control. Over the three experimental weeks, participants will undergo CGM, wearing their sensors 7 days/week. The results of this study will allow optimizing insulin therapy based on the different characteristics of pizza in patients with type 1 diabetes mellitus treated with insulin pump. This will improve glycemic control and quality of life of these patients and reduce their risk of developing chronic diabetes complications.

DETAILED DESCRIPTION:
Pizza is a typical food from Southern Italy. Its consumption is spreading worldwide. However, eating pizza is often challenging for type 1 diabetes patients due to its high glycemic index and the sustained and prolonged postprandial hyperglycaemia. Therefore, modifications of the composition and manufacturing processes able to improve the effects of pizza on postprandial blood glucose response would be well accepted.

The purpose of this study is to compare in patients with type 1 diabetes the postprandial glucose response to the consumption of three types of pizza, obtained with different leavening techniques.

Patients with type 1 diabetes treated with continuous subcutaneous insulin infusion for at least 6 months and HbA1c less than 8.0%, will be recruited at the diabetes care unit of the Federico II University teaching hospital.

The intervention will be preceded by a one-week run-in period during which participants will undergo continuous glucose monitoring (CGM) to optimize basal infusion rate and insulin-to-glycemic load ratio. Then, according to a randomized crossover design, participants will consume at home at dinner-time in random order in three different days over a 3-week period:1) a long-leavened (60 h) pizza composed of sourdough and a flour mix; 2) a short-leavened (5 h) pizza composed of sourdough and a flour mix; 3) a traditional pizza composed of brewer's yeast and refined wheat flour. Over the three experimental weeks, participants will undergo CGM, wearing their sensors 7 days/week.

The pizza- meals will be similar in energy content and macronutrient composition. The pizza dough will be prepared in a specialized factory and kept under vacuum until use. Participants will be also provided with tomato sauce and extra-virgin olive oil in the exact amount needed to prepare pizza.

The test meal will be postponed in case of premeal blood glucose levels outside the 90-150 mg/dl range or a rapid decrease/increase of glucose levels (above 1 mg/dl per min) during the previous 60 min according to CGM measurement, Pre-meal insulin doses, will be calculated based on the individual insulin-to-glycemic load ratio and will be the same on all three occasions.

At the end of the experimental period, data from CGM and insulin pump will be downloaded by dedicated informatics platforms. Participants will use the CGM system integrated with their insulin pump, i.e., the one they are accustomed to.

The primary outcome will be the postprandial blood glucose incremental area under the curve (AUC). The secondary outcomes will be blood glucose peak and time to blood glucose peak. Both primary and secondary outcomes will be evaluated by general linear model for repeated-measures ANOVA .

The results of this study will allow the optimization of insulin therapy based on the different characteristics of pizza, in patients with type 1 diabetes mellitus treated with insulin pump. This will improve glycemic control and quality of life of these patients and reduce their risk of developing chronic diabetes complications. These complications involve severe disability for patients and huge costs for the community. Moreover, considering the large consumption of pizza, the identification of changes in its composition determining a more advantageous postprandial metabolic profile could also bring benefits to the health of the general population, reducing the incidence of chronic diseases such as type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with continuous subcutaneous insulin infusion for at least 6 months
* HbA1c less than 8.0% (64 mmol/mol)

Exclusion Criteria:

* Pregnancy
* Celiac disease
* Serious microvascular and macrovascular diabetes complications including autonomic neuropathy possibly influencing gastric emptying
* Any other chronic or acute disease apart diabetes seriously affecting health status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response (AUC) | 2 hours
  Area under the curve
Postprandial glucose response (AUC) | 8 hours
  Area under the curve

SECONDARY OUTCOMES:
Blood glucose peak | 8 hours
  The maximum glucose excursion starting from the fasting values in the hours following the meal
Time to blood glucose peak | 8 hours
  The time at which the maximum glucose excursion occurred in the hours following the meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Medicine and Surgery, Naples, Italy

IPD SHARING:
Plan to Share IPD: No